CLINICAL TRIAL: NCT00173251
Title: The Difference in Presentation Level of Variant Receptors in Female Breast Tissue in Macromastia and Micromastia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9461700605
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Aging

INTERVENTIONS:
Procedure: obtain surgical specimen for analysis

SUMMARY:
There are more and more macromastic women in Taiwan, which may due to the high cholesterol foods. Patients with macromastia not only suffered from physical problems but also psychological discomforts.

DETAILED DESCRIPTION:
Large breasts cause neck and back pain, irritating grooves, cut in the skin of the shoulders by the pressure of brassiere straps, breast pain, and maceration and dermatoses in the inframammary region. From a psychological point of view, excessively large breasts can be troublesome focus of embarrassment for the teenager as well as the woman in her senior years. Unilateral hypertrophy with asymmetry heightens embarrassment. Thus, patients seek to reduce the size of their breasts.

In the human female, variant receptors were detected in epithelial cells in normal breast tissue, benign breast lesions, breast carcinoma tissue, and breast cancer cell lines2-11. The cause of the difference in breast development status is still unclear. Abnormalities at the tissue receptor level may be important in the pathophysiology of macromastia. This study aimed to make clear the difference in variant receptor levels between breast hypertrophy patients and macromastia ones by examining the receptor levels in breast tissue. Then, we could explore the possible etiology of mammary hypertrophy and macromastia.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving reduction mammoplasty

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01; Study Completion 2006-08

PRIMARY OUTCOMES:
difference in receptor expression level

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Chih Tai, M.D., Principal Investigator — National Taiwan University Hospital